CLINICAL TRIAL: NCT07135544
Title: A Single-arm, Multicenter, Exploratory Study of Adebrelimab Combined With Apatinib and Systemic Chemotherapy for Initially Unresectable Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yongjun Chen (Other)
Responsible Party: Sponsor-Investigator, Yongjun Chen, Director, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC-001
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract Cancer; Biliary Tract Cancer (CCA)
Keywords: Adebrelimab
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab combined with the GC regimen and Apatinib (Experimental): Adebrelimab 1200mg, intravenous infusion, on day 1, repeated every 3 weeks; Gemcitabine 1000mg/m2, on days 1 and 8, every 3 weeks Cisplatin 50mg/m2, on day 1, every 3 weeks Apatinib 250mg, once daily, orally
  Interventions: Drug: Adebrelimab combined with the GC regimen and Apatinib

INTERVENTIONS:
Drug: Adebrelimab combined with the GC regimen and Apatinib — Adebrelimab 1200mg, intravenous infusion, on day 1, repeated every 3 weeks; Gemcitabine 1000mg/m2, on days 1 and 8, every 3 weeks Cisplatin 50mg/m2, on day 1, every 3 weeks Apatinib 250mg, once daily, orally

SUMMARY:
This is an exploratory and prospective study, with the research subjects being patients with initially untreated and unresectable biliary tract tumors. The efficacy and safety of the treatment regimen consisting of Adebrelimab monoclonal antibody combined with targeted therapy and systemic chemotherapy were investigated.

ELIGIBILITY:
Inclusion Criteria:

- 1. Pathological or histological diagnosis of malignant tumor of the biliary tract; 2. Patients who are classified as TxNx and TxNxM1 according to the UICC/AJCC TNM staging system (9th edition, 2024), and who, based on the judgment of the research team, meet the criteria for newly diagnosed incurable cases or are not suitable for surgery; 3. Age: 18-80 years old; 4. Expected survival period > 3 months; 5. Both genders are eligible; 6. ECOG PS score of 0 or 1; 7. No severe complications, such as hypertension, coronary heart disease, and history of mental illness, no severe allergy history; non-pregnant and non-lactating; 8. The patient's organ and hematological system functions meet the following requirements:

1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
2. Platelet count ≥ 75 × 10^9/L;
3. Hemoglobin ≥ 90 g/L;
4. Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN);
5. Aspartate aminotransferase (AST) and alanine aminotransferase ≤ 2.5 x ULN;
6. Albumin ≥ 3 g/dL
7. Creatinine ≤ 1.5 x ULN 9. Patients can understand and sign the informed consent form to participate in the trial study; good compliance.

10. Newly diagnosed patients, who have not undergone any local or systemic treatment for the tumor in the past and have undergone radical resection surgery for biliary cancer, and whose disease recurs 2 years after the surgery can be included; 11. Patients with potential fertility should use a medically approved contraceptive method (such as intrauterine device, contraceptive pills, or condoms) during the study treatment and within 1 month after the end of the study treatment; and the serum or urine HCG test must be negative within 72 hours before the study enrollment, and must be non-lactating.

Exclusion Criteria:

* 1. Patients who received immune checkpoint inhibitors before enrollment, or those who directly received another stimulatory or co-inhibitory T-cell receptor (such as CTLA-4, CD137); 2. Patients who used any other investigational drug within 4 weeks before enrollment; 3. Patients with any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism after hormone replacement therapy); children with asthma who have completely recovered after adulthood and do not require any intervention can be included, but patients requiring bronchodilator drug intervention cannot be included; 4. Congenital or acquired immune deficiencies, such as infection with human immunodeficiency virus (HIV), active hepatitis B (HBV DNA > 500 IU/ml), hepatitis C (positive hepatitis C antibody, HCV-RNA above the detection limit of the analytical method), or co-infection of hepatitis B and hepatitis C; 5. Serious infections occurred within 4 weeks before the first administration (such as intravenous infusion of antibiotics, antifungal or antiviral drugs), or unexplained fever > 38.5°C during screening or before the first administration; 6. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 7. Having an uncontrolled mental disorder; 8. Concurrently having severe and/or uncontrollable diseases that may affect the participation in the study, such as unstable angina pectoris, myocardial infarction within 6 months, unstable symptomatic arrhythmia, symptomatic congestive heart failure, poorly controlled diabetes, excessive activity, uncontrollable infection after insufficient biliary drainage (such as tumor blocking the bile duct); 9. Other cancers that occurred in the past (within the past 5 years) or simultaneously, excluding non-melanoma skin cancer and carcinoma in situ; 10. History of allergy or hypersensitivity to any study drug or any monoclonal antibody; 11. Unable or unwilling to sign the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | At the end of Cycle 6 and 10 (each cycle is 21 days)
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.

SECONDARY OUTCOMES:
DCR | up to 18 months
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
PFS | up to 24 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
AE | up to 24 months
  Overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use
OS | up to 24 months
  Time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China